CLINICAL TRIAL: NCT04545229
Title: Virtual Reality Distraction to Reduce Opioid Pain Medication Use During Adult Burn Dressing Change
Brief Title: VR for Pain Management During Adult Burn Dressing Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Henry Xiang, Professor and Center Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0257
Record Dates: First submitted 2020-09-01; First posted 2020-09-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pain; Burns
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Intervention Model Description: Three-group RCT
Masking Description: In this pilot study, no masking was implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active VR-PAT (Experimental): Active VR-based Pain Alleviation Tool (VR-PAT) group played smart phone VR-PAT during the burn dressing changes.
  Interventions: Other: VR-based Pain Alleviation Tool (VR-PAT)
- Passive VR-PAT (Experimental): Passive VR-based Pain Alleviation Tool (VR-PAT) group watched smart phone VR-PAT games without interaction during the burn dressing changes.
  Interventions: Other: VR-based Pain Alleviation Tool (VR-PAT)
- Standard Care Control (No Intervention): Standard care control group used regular distraction such as background music or no distraction.

INTERVENTIONS:
Other: VR-based Pain Alleviation Tool (VR-PAT) — Four smart phone based virtual reality games developed by the Research Information Solutions and Innovation (RISI) at the Nationwide Children's Hospital.
  Arms: Active VR-PAT; Passive VR-PAT

SUMMARY:
A randomized controlled trial to evaluate the efficacy of the VR-based Pain Alleviation Tool (VR-PAT) in reducing opioid pain medication use during adult burn dressing changes.

DETAILED DESCRIPTION:
A pilot three group gender-balanced randomized clinical trial (RCT) among adult burn patients (18 years old or above) at OSU Medical Center Inpatient Burn Program. The intervention group will receive VR-PAT as a distraction tool during the dressing change procedure (active VR group) while the comparison groups will receive either a comparable passive VR distraction tool that uses the same hardware and visual/audio features, but requires no active interaction (Control Group 1), or no distraction at all (Control Group 2).

ELIGIBILITY:
Inclusion Criteria:

1. Adult burn patient age 18-70
2. First admission for acute burn requiring dressing change
3. First admission for burn injury
4. Using Opioids for dressing changes
5. Burn is ≤ 4 days post burn

Exclusion Criteria:

1. Severe burn(s) on the face/head preventing utilization of VR
2. Cognitive/motor impairment preventing valid administration of study measures
3. Unable to communicate in English
4. Prisoners and patients who were pregnant
5. Patients admitted to the ICU

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Patient self-reported pain | During burn dressing changes
  Patient self-reported pain using the 100mm Visual Analog Scale (VAS), 0 (min)-100(max), higher score for worse outcome.

SECONDARY OUTCOMES:
Opioid medication utilization, morphine equivalent dose per day during inpatient hospital stay. | Each day during inpatient hospital stays up to 7 days.
  Opioid pain medication use (converted to morphine equivalent dose), obtained through patient medical administration records. This data will be used as morphine equivalent dose per day, total morphine-equivalent dose during hospital stay, and average morphine-equivalent dose among active VR group, passive VR group, and standard care group in comparison.

OTHER OUTCOMES:
Patient VR experience | Subjective experience during burn dressing change, on average lasting 15-45 minutes.
  Patient subjective virtual reality experience using a survey questionnaire (7 items about participant's experience with VR during burning dressing changes). Questions are a mixture of yes/no and a 100 Visual Analog Scale with 0 being "Not at All" and 100 being "Very Much"
Nurse reported feasibility of VR in clinical burn wound care | Subjective observation of patient's utilization of VR during burn dressing change, on average lasting 15-45 minutes.
  Attending nurse answered two questions using a survey questionnaire about clinical feasibility of VR using scale ranging from "not at all" to "very easy".

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, Principal Investigator — The Ohio State University/Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We are not allowed to share patient medical records data.

REFERENCES:
- [Result] Armstrong M, Coffey R, Luna J, Xiang H. Pilot randomized clinical trial of virtual reality pain management during adult burn dressing changes: Lessons learned. PLOS Digit Health. 2023 Sep 25;2(9):e0000231. doi: 10.1371/journal.pdig.0000231. eCollection 2023 Sep. PMID 37747893